CLINICAL TRIAL: NCT06208709
Title: Biomechanical Treatment of CTS Via Carpal Arch Space Augmentation: A Pilot Clinical Trial
Brief Title: Carpal Arch Space Augmentation (CASA) Clinical Trial
Acronym: CASA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Zong-Ming Li, Professor, Vice Chair of Research, Department of Orthopaedic Surgery, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00003671; 1R21AR082111-01A1 (NIH)
Record Dates: First submitted 2023-12-20; First posted 2024-01-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Syndrome
Keywords: cts; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two treatment arms:
  Arm 1 - CASA device arm; Arm 2 - Standard of care (SOC) arm
  In both arms participants are being given a treatment for CTS. Throughout the intervention, participants wear their device daily while they sleep and then record their response within a daily journal. Additionally, participants are contacted weekly to answer weekly questionnaires related to their symptoms and hand function.
Who Masked: Outcomes Assessor
Masking Description: Groups in which participants are randomized into will be unknown to the investigators evaluating the outcome data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- CASA Arm (Experimental): Arm that will be given the test intervention device.
  Interventions: Device: carpal arch space augmentation (CASA)
- SOC Arm (Active Comparator): Arm that is given a standard brace used for treating Carpal Tunnel Syndrome pain.
  Interventions: Device: standard of care (SOC)

INTERVENTIONS:
Device: carpal arch space augmentation (CASA) — A BOA brace with a balloon that is affixed internally. The device applies a small cyclic force of to the wrist. The cycles include a brief period of force applied, followed by a brief period of no force. The device is intended to be worn during hours of sleep.
  Arms: CASA Arm
Device: standard of care (SOC) — A BOA brace that can be adjusted to the arm of the participant.
  Arms: SOC Arm

SUMMARY:
This research proposes to evaluate the effectiveness of a novel device designed for the treatment of carpal tunnel syndrome. The device applies a small cyclic force to the wrist. The cycles include a small time period of force is applied, followed by a brief period of no force. The device is intended to be worn during hours of sleep. The efficacy of the treatment is evaluated based on patient reported outcomes. Treatment efficacy will also be evaluated based on comparisons to patient reported outcomes for a SOC treatment.

DETAILED DESCRIPTION:
Carpal tunnel syndrome is a commonly diagnosed disorder of the hand that affects 3.7% of the population. Carpal tunnel release surgery can provide some symptomatic relief to patients but surgical transection of the transverse carpal ligament can disrupt essential anatomical, biomechanical, and physiological functions of the carpal tunnel. This clinical trial seeks to determine the effectiveness of the CASA device in alleviating CTS pain by augmenting the carpal arch space. During an early investigation of the transverse carpal ligament, investigators discovered the biomechanical mechanism of carpal arch space augmentation (CASA) for median nerve decompression. The CASA approach is supported extensively through research ﬁndings utilizing geometric modeling, ﬁnite element analysis, in vitro cadaveric experiments, and in vivo human studies.

In this proposed pilot clinical trial, investigators will compare the device's performance with a widely accepted standard of care (SOC) brace intervention (Thermoformable Exos# Wrist Brace, DJO, Vista, CA). Incorporating the CASA intervention as part of a brace is an innovative intervention study design offering a unique opportunity to identify the additive beneﬁt of CASA and for patients to beneﬁt from the combined effects of both CASA and a SOC.

This study is designed to be a randomized, single-blinded, two-arm trial. A suﬃcient number of patients will be recruited such that a total of 76 subjects will successfully complete the baseline run-in period and be randomized, with consideration of a 20% attrition rate among randomized patients, to yield 60 participants with complete data. The CASA group will be required to undergo wrist compression during the evening. The wrist compression is achieved by automated inﬂation of the balloon for a saturated pressure of 140 mmHg, which is calibrated to impart the targeted therapeutic compression force on the patient's wrist of 10 N. The intervention period will last for four weeks for the CASA group. For the SOC group, there is no compression force, as it is measuring a brace-alone condition, and will similarly last for a period of four weeks.

Patients will self-administer their assigned intervention of either CASA or sham device, and will have off-site access to study materials and questionnaire journals, thus reducing participant burden and eliminating travel expense. Data forms are designed to capture all data elements with the structure to facilitate completeness, quality, and statistical analysis. Furthermore, exploratory endpoints will be evaluated such as (a) number of participants that began to take analgesics during the study intervention phase, (b) the number of participants who opted for surgery during the intervention and post-intervention follow-up phases, (c) per-protocol comparisons of treatment arms, and (d) the impact of sex on response to treatment.

The trial will consist of 3 phases for participants; run-in, intervention, follow-up. During the run-in phase, subjects will be randomized and undergo compliance testing, along with a brief duration of device wearing, to ensure they conform with protocol instructions.

Once participants successfully complete the run-in, they will move into the intervention phase. During the intervention phase, subjects will wear their arm's respective device/brace nightly. Participants will report their adherence each day before falling asleep and once again upon waking. Participants will receive weekly phone calls in which they will report the outcome measures for the week to a member of the study team who will record the data.

After the intervention phase, participants will proceed to the follow-up phase which will last for four weeks. In this phase, participants will continue to receive weekly phone calls.

Regardless what the participant's compliance to protocol requirements for abstaining from analgesics or wearing the device 8 hours per day, the participant will be asked to complete their journals per protocol for the primary intent to treat outcome. The data gained from these patients will be used in an exploratory statistical analysis to determine if any signiﬁcant differences exist between patients who were compliant to the study and those who were not. If adherence standards are not consistently met within either treatment group, a sensitivity analysis using a per-protocol cohort will be performed. A signiﬁcance level of 0.05 will be assumed for tests of the primary outcome. Analyses of secondary outcomes will be interpreted cautiously due to multiple comparisons.

It is predicted that an intervention period of wearing the CASA device will signiﬁcantly improve patient reported outcomes of the primary endpoint, BCTQ SSS, and some of the secondary endpoints. Furthermore, it is expected that the positive effects of the CASA device intervention will continue after the treatment period has concluded. In both long-term wear and combined CASA-brace effect, it is anticipated that the CASA device group will outperform the SOC group in alleviating patient symptoms.

ELIGIBILITY:
Inclusion Criteria

* 18 and older
* Diagnosed with right-handed or bilateral CTS. Participants will be treated only in the right hand.

Exclusion Criteria

* History of musculoskeletal or neurological conditions that may confound Carpal Tunnel Syndrome symptoms, including but not limited to:

  1. Diagnosed or suspected arthritis in the test wrist, hand, or finger joints
  2. Prior neck trauma, whiplash injury, or any condition suggestive of cervical radiculopathy
  3. Current or prior treatment from a healthcare provider such as neurologist, physical therapist, physiatrist, rheumatologist, neurosurgeon, orthopedic surgeon or chiropractor for cervical radiculopathy or other musculoskeletal problem involving the neck, shoulder, and or upper extremity
* History of traumatic or chronic symptomatic neuromusculoskeletal disorders involving the upper extremity to be tested.
* The following diseases: uncontrolled diabetes, thyroid disease, rheumatoid arthritis, gout, lupus, renal failure, hemodialysis, sarcoidosis, amyloidosis, additional systemic diseases that may have an effect on the peripheral median nerve.
* Positive diagnosis of cervical disorders affecting the same side of the body as the test hand such as radiculopathy, spondylosis, tumor, and multiple sclerosis
* Symptomatic joint diseases in the test hand (e.g., Osteoarthritis)
* Osteoporosis in the test hand
* History of carpal tunnel release in the test hand
* History of corticosteroid injection treatments for CTS in the test hand within the 3 months preceding study initiation
* Women who are currently pregnant
* Patients who have carpal tunnel release surgery scheduled for the next 12 weeks in their test hand.
* Patients who have taken pain medication, including over-the-counter products, within 2 weeks prior to initiation of the study.
* Will not participate in other CTS treatment or therapies during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ SSS) | Baseline and up to 8 weeks
  The BCTQ SSS is a validated, self-reported instrument used in the assessment of pain intensity for patients with carpal tunnel syndrome. Higher numbers are worse outcomes. Possible scores range from 1 ("normal", "no pain", or "without difficulty") to 5 ("very serious", "continued", "more than 5 times")
  Change = (Baseline score - week 8 score)

SECONDARY OUTCOMES:
Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ FSS) | Baseline and up to 8 weeks
  The BCTQ FSS is a validated, self-reported instrument used in the assessment of hand function for patients with carpal tunnel syndrome. Higher numbers are worse outcomes. Possible scores range from 1 (no difficulty) to 5 (cannot perform activity at all due to symptoms)
  Change = (Baseline score - week 8 score)
Michigan Hand Outcomes Questionnaire (MHQ) | Baseline and up to 8 weeks
  The MHQ is a valid and reliable instrument for the outcomes in comparing pain and task completion between right and left hands. For scales in sections I and II of the MHQ, higher numbers are worse outcomes. Possible scores range from 1 ("very good", "not at all difficult") to 5 ("very poor", very difficult")
  For scales in sections III and IV of the MHQ, higher numbers are better outcomes. Possible scores range from 1 (always) to 5 (never).
  For scales in sections V and VI of the MHQ, higher numbers are worse outcomes. Possible scores range from 1 (strongly agree) to 5 (strongly disagree)
  Change = (Baseline score - week 8 score)
Visual Analog Scales for pain, tingling, and numbness | Baseline and up to 8 weeks
  Scales used to report pain, tingling, numbness intensity by the participant. Higher numbers are worse outcomes. Possible scores range from 0 (no pain) to 10 (worst pain).
  Change = (Baseline score - week 8 score)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
No current plan exists. If data is shared in the future, it will only be deidentified data.